CLINICAL TRIAL: NCT05795231
Title: Clinical Outcome of Endotracheal Intubation in Non-trauma Patients in the Emergency Department of Alexandria Main University Hospital
Brief Title: Clinical Outcome of Endotracheal Intubation in Non-trauma Patients
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Luther Martin Luther, Resident, Alexandria University
Other Study IDs: AlexandriaU-LutherM
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2023-03

CONDITIONS: Adverse Effects of Endotracheal Intubation
Keywords: endotracheal intubation; clinical outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Gender Based: Male patients will be compared to female patients with regards to incidence of complications
  Interventions: Device: Macintosh Laryngoscope Vs Video Laryngoscope
- Age Based: Various age groups will be evaluated to determine vulnerable age groups
  Interventions: Device: Macintosh Laryngoscope Vs Video Laryngoscope

INTERVENTIONS:
Device: Macintosh Laryngoscope Vs Video Laryngoscope — Evaluate incidence of first trial success and complications

SUMMARY:
The study will involve all adult patients visiting the Alexandria University main hospitals' Emergency department for reasons other than trauma that will require assisted ventilation via endotracheal intubation. Those pre-intubated or intubated post CPR will not be included. The main aim is to evaluate the clinical outcome (complications) of emergency endotracheal intubation and to correlate the incidence and nature of complications associated with tracheal intubations to demographic data and patient characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sex with a life threatening impairment of the cardiovascular, respiratory or neurological system requiring emergency endotracheal intubation in the emergency department of Alexandria Main University Hospital.

Exclusion Criteria:

* • Patients who are less than 18 years of age.

  * Patients intubated out of the hospital.
  * Trauma patients.
  * Patients intubated for cardiac arrest.
  * Failed intubation in the field

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the required criteria and consent to the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Major Adverse Events | 24 hours
  Severe hypoxemia, Cardiac arrest, Cardiovascular collapse, Death

SECONDARY OUTCOMES:
Moderate Complications | 24 hours
  Cardiac arrhythmia, Esophageal intubation, Aspiration, Dental injury, Difficulty intubation, Agitation

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No